CLINICAL TRIAL: NCT05923359
Title: Realtime Diagnosis From Electrocardiogram Artificial Intelligence-Guided Screening for Atrial Fibrillation With Long Follow-Up (REGAL)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Xiaoxi Yao, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-011253
Record Dates: First submitted 2023-06-19; First posted 2023-06-28 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apple Watch Intervention Group (Experimental): Participants will be asked to wear an Apple Watch and use the Mayo Clinic ECG Study App to collect and share data with the study team.
  Interventions: Other: Apple Watch
- Control Group (No Intervention): Participants will receive usual care.

INTERVENTIONS:
Other: Apple Watch — Apple Watch
  Arms: Apple Watch Intervention Group

SUMMARY:
The purpose of this research is to test whether Apple Watch, used as a long-term monitoring device, can enable early detection of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Had a 10-second 12-lead ECG done at Mayo Clinic
* Have a high AI-ECG risk score indicating a high likelihood of previously unrecognized AF
* Men with CHA2DS2-VASc2 ≥2 or women with CHA2DS2-VASc ≥ 3

Exclusion Criteria:

* Diagnosed atrial fibrillation
* Diagnosed dementia
* Diagnosed end-stage kidney disease
* History of intracranial bleeding
* Have an implantable cardiac monitoring device, including a pacemaker, a defibrillator, or implanted loop recorder
* Missing date of birth
* Residence outside of the U.S. or missing address information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation | 2 years
  Number of participants diagnosed with atrial fibrillation

SECONDARY OUTCOMES:
Change in individuals' maximum learning span | Baseline, 2 years
  Measured using the Mayo Test Drive (MTD):Test Development through Rapid Iteration, Validation and Expansion. A web-based platform for remote self-administered cognitive assessment that uses the Stricker Learning Span (SLS), which is a computer adaptive word-list memory test that matches test difficulty to user performance. Maximum learning span is total number of words recognized.
Change in processing speed measure | Baseline, 2 years
  Measured using the Mayo Test Drive (MTD):Test Development through Rapid Iteration, Validation and Expansion. A web-based platform for remote self-administered cognitive assessment that uses a symbols test to measure processing speed reported in average completion time (seconds).
Ischemic stroke or systemic embolism events | 2 years
  Number of ischemic stroke or systemic embolism events
Major bleeding | 2 years
  Number of major bleeding events
Mortality | 2 years
  Number of participant deaths

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxi Yao, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yao X, Attia ZI, Behnken EM, Hart MS, Inselman SA, Weber KC, Li F, Stricker NH, Stricker JL, Friedman PA, Noseworthy PA. Realtime Diagnosis from Electrocardiogram Artificial Intelligence-Guided Screening for Atrial Fibrillation with Long Follow-Up (REGAL): Rationale and design of a pragmatic, decentralized, randomized controlled trial. Am Heart J. 2024 Jan;267:62-69. doi: 10.1016/j.ahj.2023.10.005. Epub 2023 Oct 30. PMID 37913853
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials